CLINICAL TRIAL: NCT03434990
Title: Effects of the Spinal Manipulative Therapy and Myofascial Release on Pain Threshold, Muscle Function and Balance of Individuals With Non-specific Chronic Low Back Pain: Randomized Controlled Trial
Brief Title: Effects of the Spinal Manipulative Therapy and Myofascial Release in Individuals With Non-specific Chronic Low Back Pain
Acronym: ChiroRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Prof. Rodrigo Luiz Carregaro, Prof. Dr., University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChiroRCT
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Chronic Low Back Pain
Keywords: spinal manipulative therapy; Myofascial release; Low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal; Myofascial Release Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial, characterized by the application of manual therapy, in which subjects will be randomly allocated into two groups: spinal manipulation plus myofascial release and spinal manipulation. The participants will be individuals with non-specific chronic low back pain. The study will be reported following the recommendations of the CONSORT Statement. For the present study, non-specific chronic low back pain was defined as uninterrupted low back pain for more than 12 weeks, with unknown causes.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor won't have any knowledge about the study purposes and will be unaware of the group allocation. The statistical analysis will also be performed blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal manipulation/myofascial release (Experimental): 2x/week, for 3 weeks, performed by a chiropractor. Sessions will last 20 minutes, with 1 individual per session. Myofascial release will be done on paravertebral muscle (Erector spinae, quadratus lumborum) and on gluteus maximus and piriform muscles, the pressure will depend of pain tolerance of each subject. After this procedure, the spinal manipulation will be performed on the sacroiliac join and on the lumbar vertebrae with less mobility.
  Interventions: Other: Spinal manipulation/myofascial release
- Spinal manipulation (Active Comparator): 2x/week, for 3 weeks, performed by a chiropractor. Sessions will last 20 minutes, with 1 individual per session. The spinal manipulation will be performed on the sacroiliac join and on the lumbar vertebrae with less mobility.
  Interventions: Other: Spinal manipulation

INTERVENTIONS:
Other: Spinal manipulation/myofascial release — The protocol will be composed by myofascial release followed by spinal manipulation. Paravertebral muscles and gluteus maximus and piriform muscles will be manually checked for tension, stiffness, spasm and painful points. The intervention will be composed by: trigger points release, release of muscle fascia and active release technique. The myofacial release will be done with a constant pressure during 30 seconds, 3x in each point. After this procedure, the spinal manipulation will be performed in high velocity and low amplitude thrust technique, on the lumbar spine and sacroiliac joint.
  Other Names: Manual therapy
  Arms: Spinal manipulation/myofascial release
Other: Spinal manipulation — The sacroiliac joint will be test and manually verified for any dysfunction, and the lumbar spine will be also assessed to verify any hypomobility and vertebral rotation. The segments with alterations will be manipulated with a high velocity and low amplitude thrust technique.
  Other Names: Manual therapy
  Arms: Spinal manipulation

SUMMARY:
The aim will be to compare a experimental group submitted to a protocol of spinal manipulation and myofascial release; and a control group composed by spinal manipulation only, in individuals with chronic non-specific low back pain. This is a randomized controlled trial, characterized by the application of manual therapy, in two modalities: spinal manipulation plus myofascial release and spinal manipulation alone. Participants will be enrolled and randomly allocated into two groups: 1) spinal manipulation plus myofascial release, totaling 6 sessions, 2x/week, for 3 weeks; 2) spinal manipulation: 6 sessions, 2x/week, for 3 weeks. Participants will be evaluated in two different moments: 1) Baseline (pre-intervention); 2) at the end of intervention period (3 weeks); and 3) after 3 months follow-up. The primary outcomes will be pain intensity (measured in centimeters with the visual analogue scale - VAS) and disability (measured by the Quebec questionnaire - QDS). The secondary outcomes will be muscle fatigue (measured by the Biering-Sorensen test), postural balance (measured by the Y Balance test), pain threshold (algometry, in kgf) and perception of recovery (Likert scale of 6-points) and health status (measured by the Eq5d3L questionnaire). Data analysis will be performed with the SPSS (Statistical Package for the Social Sciences) software version 24.0. Data normality assumptions will be confirmed by the Shapiro Wilk test. If the assumptions were met, a mixed ANOVA with repeated measures will be adopted, based on the outcomes and the independent variables (groups), for the comparison between pre-intervention and post-intervention. Spinal manipulation plus myofascial release is expected to have better effects than spinal manipulation alone, associated with the outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* presence of non-specific chronic low back pain for more than 12 consecutive weeks;
* have not performed Physical Therapy, Osteopathic and/or chiropractic sessions for at least 3 months prior to the research.

Exclusion Criteria:

* history of trauma or fractures in the trunk and lumbar spine;
* presence of neural root symptoms;
* infection and inflammation on spine and upper and lower limbs for at least 3 months prior to research;
* have undergone surgery on spine, chest and abdomen;
* rheumatologic and myopathic diseases;
* renal, digestion and neurological diseases;
* use of anti-inflammatories drugs and analgesic drugs for at least 2 weeks prior the research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Change from Pre-Intervention (baseline) compared to Post-Intervention (3 weeks) and Follow up (3 months)
  Pain intensity measured by a Visual Analog Scale (in centimeters)
Disability | Change from Pre-Intervention (baseline) compared to Post-Intervention (3 weeks) and Follow up (3 months)
  Quebec Back Pain Disability Scale (scores ranging from 0 to 100)

SECONDARY OUTCOMES:
Muscle fatigue | Change from Pre-Intervention (baseline) compared to Post-Intervention (3 weeks) and Follow up (3 months)
  Muscle fatigue measured by the Biering-Sorensen test (in seconds)
Health Status | Change from Pre-Intervention (baseline) compared to Post-Intervention (3 weeks) and Follow up (3 months)
  Health Status measured by the EQ-5D-3L questionnaire, consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The responses record three levels of severity
Balance | Change from Pre-Intervention (baseline) compared to Post-Intervention (3 weeks) and Follow up (3 months)
  Y-Balance test (in cm)
Perception of Recovery | Change from Pre-Intervention (baseline) compared to Post-Intervention (3 weeks) and Follow up (3 months)
  Perception of Recovery measured by a Likert scale (6-points)
Pain threshold | Change from Pre-Intervention (baseline) compared to Post-Intervention (3 weeks) and Follow up (3 months)
  Pain threshold measured by Algometry (in kgf)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Carregaro, PhD, Principal Investigator — University of Brasilia
Locations (1):
- Complexo da Academia do Bombeiro Militar DF, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Undecided